CLINICAL TRIAL: NCT00000788
Title: A Study to Assess the Effect of Concomitant Administration of Fluconazole on the Clinical Pharmacokinetics of Methadone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: CPCRA 030; 11580 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Candidiasis; HIV Infections
Keywords: Methadone; Drug Interactions; Drug Therapy, Combination; Fluconazole; Antifungal Agents; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — Candidiasis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Methadone; Fluconazole

INTERVENTIONS:
Drug: Methadone hydrochloride
Drug: Fluconazole

SUMMARY:
To evaluate the pharmacokinetics and safety of concomitant administration of methadone and fluconazole.

Injection drug users constitute the second largest subset of the U.S. population at risk for HIV infection and AIDS-associated mortality. Narcotic addiction is often treated by use of methadone. Fluconazole has been shown to be highly effective in treating symptomatic mucosal candidiasis, but it is unknown whether fluconazole affects methadone metabolism, which could result in symptoms of methadone withdrawal or overdose in patients taking the drugs in combination.

DETAILED DESCRIPTION:
Injection drug users constitute the second largest subset of the U.S. population at risk for HIV infection and AIDS-associated mortality. Narcotic addiction is often treated by use of methadone. Fluconazole has been shown to be highly effective in treating symptomatic mucosal candidiasis, but it is unknown whether fluconazole affects methadone metabolism, which could result in symptoms of methadone withdrawal or overdose in patients taking the drugs in combination.

Patients are randomized to receive methadone plus either fluconazole or placebo in clinic daily for 16 days. Study drugs are administered as close to 8 AM as possible. Patients must visit the Fort Greene clinic on study days 1, 2, 15, and 16; they may receive treatment at their home clinics on days 3 through 14.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy.
* Intermittent acetaminophen, aspirin, and ibuprofen.

Patients must have:

* CD4 count >= 250 cells/mm3 within 3 months prior to study entry.
* Received a stable dose of methadone for a minimum of 30 days prior to study entry.
* Negative urine toxicology screen (except for methadone or methadone metabolites) within 14 days prior to study entry.
* Reasonably good health.
* Life expectancy of at least 6 months.
* Ability and willingness to comply with protocol requirements.

NOTE:

* Patients will be recruited from the methadone maintenance treatment program currently administered by Addiction Research and Treatment Corporation. Enrollment of women is encouraged.

NOTE:

* Patients who are currently enrolled in CPCRA treatment and prophylaxis trials are eligible for this study provided they have been permanently removed from study drug on the other protocol.

Prior Medication:

Required:

* Stable dose of methadone for a minimum of 30 days prior to study entry.

Allowed:

* Prior antiretroviral therapy (dose should be stable for 14 days prior to study entry).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known sensitivity to azoles, methadone, and other opiate narcotics.

Concurrent Medication:

Excluded:

* Amiodarone.
* Anesthetics, general.
* Barbiturates.
* Carbamazepine.
* Cimetidine.
* Ciprofloxacin.
* Dexamethasone.
* Disulfiram.
* Erythromycin.
* Fluoroquinolones.
* Fluoxetine.
* Gestodene.
* Hydrochlorothiazide.
* Hypoglycemics, oral.
* Isoniazid.
* Itraconazole.
* Ketoconazole.
* Levomepromazine.
* MAO inhibitors.
* Methoxsalen.
* Nafcillin.
* Narcotic analgesics.
* Naringenin.
* Norethindrone.
* Omeprazole.
* Pentazocine.
* Phenothiazines.
* Phenytoin.
* Quinidine.
* Ranitidine.
* Rifabutin.
* Rifampin.
* Sedative hypnotics.
* Sulfaphenazole.
* Tranquilizers.
* Tricyclic antidepressants.
* Troleandomycin.
* Warfarin.

Prior Medication:

Excluded within 30 days prior to study entry:

* Ketoconazole, fluconazole, or itraconazole.
* Experimental drugs.

Alcohol or illicit drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Study Completion 1994-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cobb M, Study Chair; Letts A, Study Chair
Locations (1):
- Addiction Research and Treatment Corp, Brooklyn, New York, United States

REFERENCES:
- [Background] Cobb MN, Desai J, Brown LS Jr, Zannikos PN, Rainey PM. The effect of fluconazole on the clinical pharmacokinetics of methadone. Clin Pharmacol Ther. 1998 Jun;63(6):655-62. doi: 10.1016/S0009-9236(98)90089-3. PMID 9663180